CLINICAL TRIAL: NCT03282474
Title: HepNet Pilot Trial: Multicenter Trial for the Treatment of Chronic Hepatitis E With Sofosbuvir (SofE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: HepNet Study House, German Liverfoundation (Network); Gilead Sciences (Industry); German Center for Infection Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HepNet-SofE; 2017-000403-24 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis E; Hepatitis Chronic Viral
Keywords: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — Sofosbuvir

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm multicenter, phase II pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sofosbuvir (Experimental): Sofosbuvir 400 MG film-coated tablet, oral administration of one tablet once daily for 24 weeks.
  Interventions: Drug: Sofosbuvir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 MG Oral Tablet [Sovaldi]
  Other Names: Sovaldi

SUMMARY:
This is a single arm multicenter pilot study to provide preliminary evidence whether sofosbuvir (SOF) is efficacious and can be safely used in patients with chronic Hepatitis E virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥ 18 years
3. Confirmation of chronic HEV infection documented by: Positive HEV RNA at least 3 months before Screening, and positive for HEV RNA at the time of Screening
4. Documented previous ribavirin therapy or documented contraindication for full dose (≥ 600mg qd) ribavirin monotherapy for at least 3 months
5. Body mass index (BMI) ≥ 18 kg/m2
6. Screening ECG without clinically significant abnormalities
7. Subjects must have the following laboratory parameters at screening:

   * Platelets ≥ 60,000/μL
   * INR ≤2.0 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * HbA1c ≤ 10%
   * Creatinine clearance (CLcr) ≥ 30 mL/min, as calculated by the Cockcroft-Gault equation (using actual body weight)
8. Subject has not been treated with any investigational drug or device within 42 days of the Screening visit
9. A negative serum pregnancy test is required for female subjects (unless surgically sterile or women ≥ 54 years of age with cessation for 24 ≥ months of previously occurring menses).

   Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

   Or

   Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from the date of Screening until 30 days after last dose of study drug:
   * intrauterine device (IUD) with a failure rate of < 1% per year
   * female barrier method: cervical cap or diaphragm with spermicidal agent
   * tubal sterilization
   * vasectomy in male partner
   * hormone-containing contraceptive:

     * implants of levonorgestrel
     * injectable progesterone
     * oral contraceptives (either combined or progesterone only)
     * contraceptive vaginal ring
     * transdermal contraceptive patch
10. Subject must be able to comply with the dosing instructions for study drug administration and be able to complete the study schedule of assessments.

Exclusion Criteria:

1. Clinically-significant illness (other than HEV) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol.
2. Ribavirin administration within the last 28 days.
3. Infection with the hepatitis C virus (defined as HCV RNA positive)
4. Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug (for example, gastric bypass or severe ulcerative colitis).
5. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
6. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 2 years. Subjects with psychiatric illness that is wellcontrolled on a stable treatment regimen for at least 12 months prior to screening or has not required medication in the last 12 months may be included.
7. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
8. Pregnant or nursing female
9. Clinically-relevant drug or alcohol abuse within 12 months of screening including any uncontrolled drug use within 6 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the investigator. Uncontrolled users of intravenous drugs will not be permitted to enroll in the study.
10. Use of any prohibited concomitant medications within 21 days of the Baseline/Day 1 visit.

    Use of Amiodaron as concomitant medication is prohibited within 60 days of Baseline/Day1 visit.
11. Known hypersensitivity to SOF or formulation excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who become HEV RNA negative after 24 weeks of therapy | after 24 weeks of therapy
  Measured by the proportion of subjects who become HEV RNA negative (HEV RNA undetectable)

SECONDARY OUTCOMES:
Proportion of subjects who are HEV RNA negative 12 weeks after discontinuation of therapy | 12 weeks after discontinuation of therapy (week 36)
  Viral load measurement
Additional efficacy evaluations include HEV RNA change from baseline during therapy | after 2 days, 4 days, 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks,16 weeks, 20 weeks, and 24 weeks of therapy
  Viral load and laboratory measurements
Comparison of proportion of patients who are HEV RNA negative after rapid or slow decline of HEV viral load after 24 weeks of therapy | after 24 weeks of therapy
  Viral load measurement
Proportion of subject who reached ALT normalization after 12 weeks and 24 weeks of therapy and 12 weeks after discontinuation of therapy | after 12 and 24 weeks of therapy and 12 weeks after discontinuation of therapy (week 36)
  Laboratory measurement
Assessment of safety: Adverse events and safety laboratory tests will be collected throughout the study | through study completion, an average of 36 weeks
  Collection of adverse events and safety laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Markus Cornberg, Prof. Dr., Principal Investigator — Hannover Medical School, Clinic for Gastroenterology, Hepatology, and Endocrinology
Locations (3):
- Germany (3):
  - Hannover Medical School, Clinic for Gastroenterology, Hepatology, and Endocrinology, Hanover, Lower Saxony
  - Charité, Campus Virchow-Klinikum, Medical Department, Division of Hepatology and Gastroenterology, Berlin
  - University Medical Center Hamburg-Eppendorf, Center for Internal Medicine, I. Medical Clinic and Polyclinic, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahid A, Meyer N, Wundes C, Huffner L, Janshoff S, Frericks N, Friesland M, Dinkelborg K, Aliabadi E, Laue F, Cornberg M, Maasoumy B, Bremer B, Pischke S, Muller T, Wiesch JZS, Benckert J, Ulrich RG, Hardtke S, Dorge P, Vondran F, Lohse A, Manns MP, Todt D, Wedemeyer H, Pietschmann T, Steinmann E, Gomer A, Behrendt P. Extrahepatic Replication and Genomic Signatures of the Hepatitis E Virus in the Kidney. Liver Int. 2025 Jul;45(7):e70183. doi: 10.1111/liv.70183. PMID 40575997
- [Derived] Gomer A, Klohn M, Jagst M, Nocke MK, Pischke S, Horvatits T, Schulze Zur Wiesch J, Muller T, Hardtke S, Cornberg M, Wedemeyer H, Behrendt P, Steinmann E, Todt D. Emergence of resistance-associated variants during sofosbuvir treatment in chronically infected hepatitis E patients. Hepatology. 2023 Dec 1;78(6):1882-1895. doi: 10.1097/HEP.0000000000000514. Epub 2023 Jun 20. PMID 37334496
- [Derived] Cornberg M, Pischke S, Muller T, Behrendt P, Piecha F, Benckert J, Todt D, Steinmann E, Papkalla A, von Karpowitz M, Koch A, Lohse A, Hardtke S, Manns MP, Wedemeyer H. Sofosbuvir monotherapy fails to achieve HEV RNA elimination in patients with chronic hepatitis E - The HepNet SofE pilot study. J Hepatol. 2020 Sep;73(3):696-699. doi: 10.1016/j.jhep.2020.05.020. Epub 2020 Jul 2. No abstract available. PMID 32624195